CLINICAL TRIAL: NCT04784221
Title: Nanoparticles and Hypofractionated Protontherapy for Reirradiation of Pantumor Relapse: NANOPRO, a Non-randomized Phase II Study
Brief Title: Nanoparticles and Hypofractionated Protontherapy for Reirradiation of Pantumor Relapse
Acronym: NANOPRO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study prematurely terminated following the decision by industrial partner to withdraw from the project (product supply issue).
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003671-17
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Cancer; Previous Radiation
Keywords: protontherapy; nanoparticles; AguIX
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation by protontherapy associated to nanoparticles injection (Experimental)
  Interventions: Radiation: Radiation by protontherapy associated to nanoparticles injection

INTERVENTIONS:
Radiation: Radiation by protontherapy associated to nanoparticles injection — Treatment for the study will be based on proton therapy and the administration of AGuIX® nanoparticles.
  Protontherapy will be carried out for 4 consecutive weeks with 5 sessions per week (20 sessions) from D1 to D26.
  The administration of the AGuIX® nanoparticle will be done on Days 1, 8 and 15 during protontherapy

SUMMARY:
This is a prospective multicenter non-randomized phase II study: proton therapy with nanoparticles based on polysiloxane and gadolinium chelates injectable intravenously

DETAILED DESCRIPTION:
This is a prospective multicenter non-randomized phase II study: proton therapy with nanoparticles based on polysiloxane and gadolinium chelates injectable intravenously in recurrent tumors

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Patient with tumor of the cephalo-spino-iliosacral axis corresponding to the spectrum of tumors treated in protontherapy, particularly base of the skull, pharyngeal wall, parapharyngeal and retropharyngeal lymph nodes, cavum without associated lymph node, pre-spinal tumor, etc. tumors are immobile as opposed to visceral thoracic, abdominal and pelvic tumors which may be mobile which will be excluded because they cannot be irradiated in proton therapy in the current state of the art),
* Tumor already irradiated, within more than 6 months before inclusion
* Patient with a relapse or a new tumor in irradiated territory
* Tumor considered to be radioresistant (TCD50> 50Gy)
* Dosimetry (s) of previous irradiations available
* Progressive tumor in tissue already irradiated to at least 40 Gy EQD2 (α / β = 2)
* Indication of reirradiation by protontherapy for curative purposes. The indication for reirradiation by protontherapy will be discussed depending on the size and location of the tumor (particularlyfor a volume of less than or equal to 113 ml of PTV in an ENT situation may be taken into account), the presence of previous toxicities. It will be validated by RCP at the Center François Baclesse
* The patient may have received previous systemic treatment
* Evaluable disease according to RECIST 1.1 criteria
* Performance Status ≤ 2
* Normal renal function: creatinine clearance ≥ 50 ml / min
* Patient affiliated to a social security system
* Patient having given written consent

Exclusion Criteria:

* Mobile tumors
* Lymphomas, brain tumors (gliomas), meningiomas, skin carcinomas, malignant melanomas (skin or mucous membranes), tumor of the larynx, mobile lesions of the oral cavity
* Recurrence occurring within 6 months of the end of the first irradiation
* Patient with a contraindication to radiotherapy
* Patient with progressive visceral or cerebral metastases
* Life-threatening comorbidities within two years
* Patient with a contraindication to MRI
* Immovable metallic material in the target volume (significant imaging artefacts)
* Impossibility of completely immobilizing the target volume (moving organ)
* Large volume to be irradiated (PTV) for an acceptable benefit / risk balance evaluated in RCP of the François Baclesse Center
* Neoplasic skin ulceration
* Doses previously received by OARs or radiation toxicity already present preventing reirradiation including in protontherapy (clinical and dosimetric study of each case)
* Concomitant cancer treatment such as chemotherapy, immunotherapy, targeted therapy or other, underway or planned to be initiated during irradiation
* Simultaneous participation in another therapeutic clinical trial
* Patient deprived of liberty, under guardianship or curatorship
* Pregnant or breastfeeding patient
* Patient unable to undergo medical monitoring of the trial for geographic, social or psychopathological reasons
* History of other malignant disease in the past 3 years, except skin cancer other than melanoma, carcinoma in situ of the cervix. Any other solid tumor or lymphoma (without bone marrow involvement) must have been treated and not show signs of recurrence for at least 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Local efficacy of a treatment combining the administration of nanoparticles with proton therapy | 2 years after the treatment
  proportion of patients alive and without local progression two years after the start of proton therapy (local progression-free survival rate)

IPD SHARING:
Plan to Share IPD: No